CLINICAL TRIAL: NCT01211028
Title: Safety of Autologous Adipose Derived Stroma/Stem Cells to Treat Critical Leg Ischemia.
Brief Title: Adipose CELL Derived Regenerative Endothelial Angiogenic Medicine
Acronym: ACELLDREAM
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Collaborators: French Blood Establishment (Other); Clinical Research Center, Toulouse (Other); Centre National de la Recherche Scientifique, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0405402
Record Dates: First submitted 2010-03-31; First posted 2010-09-29 (Estimated); Last update posted 2017-05-11 (Actual); Status verified 2017-05

CONDITIONS: Peripheral Vascular Diseases; Cardiovascular Diseases
Keywords: Critical leg ischemia; Adipose derived Stroma/Stem Cells; Autologous; Angiogenesis
MeSH Terms: conditions — Peripheral Vascular Diseases; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Autologous ASCs (Other): Expanded autologous ASCs (Adipose Stroma/Stem Cells) Intramuscular dose of 100 million expanded cells.
  Interventions: Biological: Expanded autologous ASCs

INTERVENTIONS:
Biological: Expanded autologous ASCs — Drug: Expanded autologous adipose-derived adult stroma/stem cells
  Other Names: Expanded autologous Adipose-derived adult Stroma/Stem cells

SUMMARY:
The main purpose of this study is to evaluate the safety and feasibility of regenerative therapy with expanded adipose derived stroma/stem cells sue, administered intramuscularly in patients with critical leg ischemia.

ELIGIBILITY:
Inclusion Criteria:

* Severe peripheral vascular disease not amenable to bypass or angioplasty
* Age >40 years old
* Normal renal function (creatinine < 1.6)
* Non pregnant female
* Lifespan > 6 months

Exclusion Criteria:

* Age <40 years old
* Refusal to give informed consent and/orCognitively disabled
* Congestive heart failure or stroke in the last 3 months
* History of cancer or myeloproliferative disorders
* Proliferative retinopathy
* Pregnancy
* Positive screening test for HIV, Hepatitis B or Hepatitis C
* Buerger patient
* Cachexia or predicted impossibility for a biopsy of at least 30 grams of fat tissue
* Pregnancy or lactation
* Having been non controlled severe pathology

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2009-01; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Number and Nature of Adverse Events : safety and tolerability | 15 days, 1, 2, 3, 4,5, 6 months for adverse events record
  To evaluate safety and tolerability related to the intramuscular injection of autologous adipose derived stroma/ stem cells. [ Designated as safety issue: Yes ]

CONTACTS AND LOCATIONS:
Overall Officials: Alessandra BURA-RIVIERE, Pr, Principal Investigator — University Hospital of Toulouse, Rangueil
Locations (1):
- University Hospital of Toulouse, Rangueil, Toulouse, France

REFERENCES:
- [Background] Planat-Benard V, Silvestre JS, Cousin B, Andre M, Nibbelink M, Tamarat R, Clergue M, Manneville C, Saillan-Barreau C, Duriez M, Tedgui A, Levy B, Penicaud L, Casteilla L. Plasticity of human adipose lineage cells toward endothelial cells: physiological and therapeutic perspectives. Circulation. 2004 Feb 10;109(5):656-63. doi: 10.1161/01.CIR.0000114522.38265.61. Epub 2004 Jan 20. PMID 14734516